CLINICAL TRIAL: NCT03011346
Title: Safety and Efficacy of the Symetis ACURATE Neo/TF Compared to the Edwards SAPIEN 3 Bioprosthesis for Transcatheter Aortic Valve Implantation by Transfemoral Approach.
Brief Title: Safety and Efficacy of the Symetis ACURATE Neo/TF Compared to the Edwards SAPIEN 3 Bioprosthesis.
Acronym: SCOPE I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V 4.0, 13.08.2018
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve stenosis; Transcatheter aortic valve implantation; Transcatheter aortic valve replacement; Randomized controlled trial
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symetis ACURATE neo/TF transfemoral TAVI system (Active Comparator): Symetis ACURATE neo/TF transfemoral TAVI system: self-expandable transcatheter aortic bioprosthesis, support frame made of nitinol, supra-annular processed trileaflet porcine pericardial valve and an outer skirt to mitigate paravalvular regurgitation (manufactured by Symetis SA, Ecublens, Switzerland)
  Interventions: Device: Symetis ACURATE neo/TF transfemoral TAVI system
- Edwards Sapien 3 Transcatheter Heart Valve (Active Comparator): Edwards SAPIEN 3 Transcatheter Heart Valve system: balloon-expandable transcatheter aortic bioprosthesis, support frame made of cobalt-chromium, three leaflets constructed of processed bovine pericardial tissue and an outer polyethylene terephthalate (PET) sealing cuff to mitigate paravalvular regurgitation (manufactured by Edwards Lifesciences, Inc., Irvine, California, USA)
  Interventions: Device: Edwards Sapien 3 Transcatheter Heart Valve

INTERVENTIONS:
Device: Symetis ACURATE neo/TF transfemoral TAVI system — Transcatheter aortic valve implantation of a Symetis ACURATE neo/TF bioprosthesis by transfemoral access, pre-dilatation mandatory.
  Arms: Symetis ACURATE neo/TF transfemoral TAVI system
Device: Edwards Sapien 3 Transcatheter Heart Valve — Transcatheter aortic valve implantation of an Edwards Sapien 3 bioprosthesis by transfemoral access.
  Arms: Edwards Sapien 3 Transcatheter Heart Valve

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is an established treatment option for patients with severe symptomatic aortic stenosis and at increased risk for surgical aortic valve replacement (SAVR). Many novel devices are currently being developed and established transcatheter heart valves undergo design reiterations to address limitations and reduce complication rates associated with the device and implantation procedure. However, device comparisons by use of randomized trials are scarce in particular for newer generation transcatheter valves. The aim of this study is to assess non-inferiority of the self-expandable Symetis ACURATE neo/TF in comparison to the balloon-expandable Edwards SAPIEN 3 transcatheter aortic valve bioprosthesis with regard to early safety and clinical efficacy at 30 days.

DETAILED DESCRIPTION:
Background:

Transcatheter aortic valve implantation (TAVI) is an established and valuable treatment option for patients with severe symptomatic aortic stenosis and at increased risk for surgical aortic valve replacement (SAVR). The use of TAVI is rapidly expanding worldwide and the indications for TAVI are widening into lower risk populations in view of favorable outcomes among high and intermediate risk patients. Many novel devices are currently developed or established devices undergo design reiterations to address limitations, such as vascular access complications, paravalvular regurgitation, and atrio-ventricular conductance disturbances. However, device comparisons by use of randomized trials are scarce in particular for newer generation transcatheter valves.

The Symetis ACURATE neo/TF, a self-expandable transcatheter valve delivered via transfemoral access, gained Conformité Européenne (CE) marking in September 2014 after showing favorable procedural and short term results. The SCOPE I trial will compare its performance to the balloon-expandable Edwards SAPIEN 3, a widely used and well-established transcatheter heart valve of the second generation, in a randomized fashion.

Objectives:

The primary objective is the comparison of the Symetis ACURATE neo/TF to the Edwards SAPIEN 3 transcatheter aortic bioprosthesis with regard to early safety and clinical efficacy at 30 days. Secondary objectives involve the comparison between the two devices with regard to secondary clinical and echocardiographic endpoints at 30 days, 1 year and 3 years.

Methods:

Sample Size: Based on an anticipated incidence proportion of 22% for the primary non-hierarchical composite endpoint at 30 days in both treatment arms, a non-inferiority margin of 7.7%, a power of 80%, a one-tailed significance level of α = 0.05, and a low attrition rate, the total required sample size amounts to 730 patients.

Design: Patients will be allocated to the Symetis ACURATE neo/TF or the Edwards SAPIEN 3 bioprosthesis at a 1:1 ratio by means of a randomly permuted block randomisation stratified on study center and Society of Thoracic Surgeons' predicted risk of mortality score (STS-PROM) strata (< 3%, ≥ 3 to < 8%, ≥ 8%).

Analysis: Estimates of the risk-differences between the two treatment arms with regard to the primary endpoint will be pooled over the predefined STS-PROM strata by means of the Cochran-Mantel-Haenszel method and Wald-type confidence limits will be calculated using the Sato variance estimator. The non-inferiority assumption will be tested at a one-sided significance level with a type I error rate (α) = 0.05. The analysis of the primary composite endpoint will be conducted according to the intention-to-treat (ITT) and the per protocol (PP) principle and non-inferiority should be claimed only if met by both.

In case non-inferiority is established, a superiority analysis will be performed using a two-tailed significance level with a type I error rate of α = 0.05. Further secondary analyses will evaluate between group differences in relation to demographic, clinical, procedural, functional and imaging characteristics. Pre-specified subgroup analyses will be conducted by use of appropriate interaction tests contrasting categories of sex, STS-PROM score (< 3%, ≥ 3 to < 8%, ≥ 8%), left ventricular ejection fraction (< 50% vs. ≥ 50%), and native aortic valve eccentricity index (≤ 0.25 vs. > 0.25).

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe aortic stenosis defined by an aortic valve area (AVA) < 1cm2 or AVA indexed to body surface area (BSA) of < 0.6 cm2/m2, including low-flow severe aortic stenosis defined by stroke volume index (SVI) < 35ml/m2, as assessed by integration of echocardiographic and invasive measurements
* Subject is symptomatic (heart failure symptoms with New York Heart Association (NYHA) Functional Class > I, angina or syncope)
* Patient is considered at increased risk for mortality if undergoing conventional surgical aortic valve replacement or judged as not operable as determined either

  * by a Logistic EuroSCORE > 20 % OR
  * by a STS-PROM score > 10% OR
  * by the heart team consisting of at least one cardiologist and cardiac surgeon based on the integration of individual clinical and anatomical factors not captured by risk-scores, the patient's age, frailty and life-expectancy
* The heart team agrees on eligibility of the patient for participation and that TAVI by transfemoral access constitutes the most appropriate treatment modality, from which the patient will likely benefit most
* Aortic annulus dimensions suitable for both valve types (area range: 338-573 mm2 AND perimeter range: 66-85 mm) based on ECG-gated multislice computed tomographic measurements. Findings of transesophageal echocardiography (TEE) and conventional aortography should be integrated in the anatomic assessment if available
* Arterial aorto-iliac-femoral axis suitable for transfemoral access with a minimum access vessel diameter ≥ 6 mm as assessed by multislice computed tomographic angiography and/or conventional angiography
* Written informed consent of the patient or her/his legal representative
* Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up

Exclusion Criteria:

* Non-valvular aortic stenosis
* Congenital aortic stenosis or unicuspid or bicuspid aortic valve
* Non-calcific acquired aortic stenosis
* Anatomy not appropriate for transfemoral transcatheter aortic valve implantation due to size of the aortic annulus or degree or eccentricity of calcification of the native aortic valve or tortuosity of the aorta or ilio-femoral arteries
* Emergency procedure including patients in cardiogenic shock (low cardiac output, vasopressor dependence, mechanical hemodynamic support)
* Severely reduced left ventricular (LV) function (ejection fraction < 20%)
* Pre-existing prosthetic heart valve in aortic position
* Presence of mitral valve prosthesis
* Concomitant planned procedure except for percutaneous coronary intervention (PCI)
* Planned non-cardiac surgery within 30 days
* Stroke within 30 days of the procedure.
* Myocardial infarction within 30 days of the procedure (except type 2)
* Evidence of intra-cardiac mass, thrombus or vegetation
* Severe coagulation conditions
* Inability to tolerate anticoagulation/anti-platelet therapy
* Active bacterial endocarditis or other active infections
* Hypertrophic cardiomyopathy with or without obstruction
* Contraindication to contrast media or allergy to nitinol
* Participation in another trial, which would lead to deviations in the preparation or performance of the intervention or the post-implantation management from this protocol

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 739 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Modified* combined early safety and clinical efficacy as defined by the Valve Academic Research Consortium-2 (VARC-2) | 30 days
  (* "NYHA class III or IV" is omitted due to lack of objectiveness in its ascertainment)
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening or disabling bleeding
  * Acute kidney injury (stage 2 or 3, including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve related dysfunction requiring repeat procedure (balloon aortic valvuloplasty, TAVI or SAVR in a separate intervention)
  * Rehospitalization for valve-related symptoms or worsening congestive heart failure
  * Valve-related dysfunction: prosthetic aortic valve stenosis (mean gradient ≥ 20 mmHg, effective orifice area ≤ 0.9-1.1cm2 and/or Doppler velocity index < 0.35) AND/OR ≥ moderate prosthetic valve regurgitation)

SECONDARY OUTCOMES:
Device success | 30 days
  Combined endpoint composed of:
  * Absence of procedural mortality AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, AND no moderate or severe prosthetic valve regurgitation)
Early safety | 30 days
  Combined endpoint composed of:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening or disabling bleeding
  * Acute kidney injury - stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (balloon aortic valvuloplasty, TAVI, or SAVR)
Clinical efficacy | 30 days
  Combined endpoint composed of:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Requiring hospitalizations for valve-related symptoms or worsening congestive heart failure
  * NYHA class III or IV
  * Valve-related dysfunction (mean aortic valve gradient ≥ 20 mmHg, effective orifice area (EOA) ≤ 0.9-1.1 cm2 and/or Doppler velocity index (DVI) < 0. 35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
Time-related valve safety | 30 days, 1 year
  Combined endpoint composed of:
  * Structural valve deterioration (Valve-related dysfunction (mean aortic valve gradient ≥ 20 mmHg, EOA ≤ 0.9-1.1 cm2 (depending on body surface area (BSA)) and/or DVI < 0.35 m/s AND/OR moderate or severe prosthetic valve regurgitation)) OR Requiring repeat procedure (TAVI or SAVR)
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thrombo-embolic events (e.g. stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy (e.g. trauma)
All-cause mortality | 30 days, 1 year, 3 years
All stroke (disabling and non-disabling) | 30 days, 1 year, 3 years
Life-threatening or disabling bleeding | 30 days, 1 year, 3 years
  * Fatal bleeding (Bleeding Academic Research Consortium (BARC) type 5)OR
  * Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC type 3b and 3c) OR
  * Bleeding causing hypovolaemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b) OR
  * Overt source of bleeding with drop in haemoglobin ≥5 g/dL or whole blood or packed red blood cells (RBCs) transfusion ≥4 units (BARC type 3b)
Acute kidney injury (stage 2 or 3, including renal replacement therapy) | 30 days, 1 year, 3 years
  * Stage 2: Increase in serum creatinine to 200-299% (2.0-2.99 × increase compared with baseline) OR Urine output <0.5 mL/kg/h for >12 but <24 h
  * Stage 3: Increase in serum creatinine to ≥300% (>3 × increase compared with baseline) OR serum creatinine of ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L) OR Urine output <0.3 ml/kg/h for ≥24 h OR Anuria for ≥12 h Notes: The increase in creatinine must occur within 48 h. Patients receiving renal replacement therapy are considered to meet Stage 3 criteria irrespective of other criteria.
Coronary artery obstruction requiring intervention | 30 days, 1 year, 3 years
Major vascular complication | 30 days, 1 year, 3 years
  * Aortic dissection, aortic rupture, annulus rupture, left ventricle perforation, or new apical aneurysm/pseudo-aneurysm OR
  * Access-related vascular injury (dissection, stenosis, perforation, rupture, arterio-venous fistula, pseudoaneurysm, haematoma, irreversible nerve injury, compartment syndrome, percutaneous closure device failure) leading to death, life-threatening or major bleeding, visceral ischaemia, or neurological impairment OR
  * Distal embolization (non-cerebral) from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage OR
  * Use of unplanned endovascular or surgical intervention associated with death, major bleeding, visceral ischaemia or neurological impairment OR
  * Any new ipsilateral lower extremity ischaemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram OR
  * Surgery for access site-related nerve injury OR
  * Permanent access site-related nerve injury
Valve related dysfunction requiring repeat procedure (balloon aortic valvuloplasty, TAVI or SAVR in a separate intervention) | 30 days, 1 year, 3 years
Rehospitalization for valve-related symptoms or worsening congestive heart failure | 30 days, 1 year, 3 years
Valve-related dysfunction: prosthetic aortic valve stenosis AND/OR ≥ moderate prosthetic valve regurgitation | 30 days, 1 year, 3 years
  Prosthetic aortic valve stenosis: mean gradient ≥ 20 mmHg, EOA ≤ 0.9-1.1cm2 and/or DVI < 0.35)
Conversion to open heart surgery | procedural
Annular rupture | procedural
New pacemaker implantation | 30 days, 1 year, 3 years
Valve thrombosis | 30 days, 1 year, 3 years
  Any thrombus attached to or near an implanted valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment. Note that valve-associated thrombus identified at autopsy in a patient whose cause of death was not valve-related should not be reported as valve thrombosis.
Mean trans-prosthetic aortic gradient | 30 days, 1 year, 3 years
Aortic regurgitation | 30 days, 1 year, 3 years
Kansas City Cardiomyopathy Questionnaire (KCCQ)-12 score | 30 days, 1 year, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pigrim, Prof. MD, Principal Investigator — Bern University Hospital, Dep. of Cardiology, 3010 Bern, Switzerland
Locations (20):
- Germany (15):
  - Herz- und Gefäss-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale, Bad Neustadt
  - Klinkum Augsburg, Augsburg
  - Zentralklinik Bad Berka, Bad Berka
  - Herz- und Gefässzentrum Bad Beversen, Bad Bevensen
  - Kerckhoff-Klinik, Bad Nauheim
  - Herzzentrum Uniklinik Köln, Cologne
  - St.-Johannes-Hospital, Dortmund
  - Herzzentrum Dresden, Dresden
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - ViDia Kliniken, Karlsruhe
  - Klinik für Herzchirurgie Karlsruhe, Karlsruhe
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum München, München
  - Klinik und Poliklinik für Herz-, Thorax- und herznahe Gefäßchirurgie, Regensburg
- University Medical Center Utrecht, Utrecht, Netherlands
- Switzerland (3):
  - Bern University Hospital, Bern
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lanz J, Kim WK, Walther T, Burgdorf C, Mollmann H, Linke A, Redwood S, Thilo C, Hilker M, Joner M, Thiele H, Conzelmann L, Conradi L, Kerber S, Schymik G, Prendergast B, Husser O, Stortecky S, Heg D, Juni P, Windecker S, Pilgrim T; SCOPE I investigators. Safety and efficacy of a self-expanding versus a balloon-expandable bioprosthesis for transcatheter aortic valve replacement in patients with symptomatic severe aortic stenosis: a randomised non-inferiority trial. Lancet. 2019 Nov 2;394(10209):1619-1628. doi: 10.1016/S0140-6736(19)32220-2. Epub 2019 Sep 27. PMID 31570258
- [Derived] Tomii D, Lanz J, Thiele H, Heg D, Kim WK, Joner M, Mollmann H, Burgdorf C, Linke A, Redwood S, Hilker M, Conradi L, Kerber S, Thilo C, Toggweiler S, Walther T, Prendergast B, Windecker S, Pilgrim T. Obstructive Coronary Artery Disease and Health Status in Transcatheter Aortic Valve Replacement: A Post Hoc Analysis of the SCOPE I Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2547111. doi: 10.1001/jamanetworkopen.2025.47111. PMID 41364435
- [Derived] Lanz J, Mollmann H, Kim WK, Burgdorf C, Linke A, Redwood S, Hilker M, Joner M, Thiele H, Conzelmann L, Conradi L, Kerber S, Thilo C, Toggweiler S, Prendergast B, Husser O, Stortecky S, Deckarm S, Kunzi A, Heg D, Walther T, Windecker S, Pilgrim T; SCOPE I Investigators. Final 3-Year Outcomes of a Randomized Trial Comparing a Self-Expanding to a Balloon-Expandable Transcatheter Aortic Valve. Circ Cardiovasc Interv. 2023 Jul;16(7):e012873. doi: 10.1161/CIRCINTERVENTIONS.123.012873. Epub 2023 Jul 7. PMID 37417229
- [Derived] Kim WK, Walther T, Burgdorf C, Mollmann H, Linke A, Redwood S, Thilo C, Hilker M, Joner M, Thiele H, Conzelmann L, Conradi L, Kerber S, Schymik G, Prendergast B, Husser O, Blumenstein J, Stortecky S, Heg D, Kunzi A, Juni P, Windecker S, Pilgrim T, Lanz J; SCOPE I Investigators. One-Year Outcomes of a Randomized Trial Comparing a Self-Expanding With a Balloon-Expandable Transcatheter Aortic Valve. Circulation. 2021 Mar 23;143(12):1267-1269. doi: 10.1161/CIRCULATIONAHA.120.052251. Epub 2021 Mar 22. No abstract available. PMID 33750210